CLINICAL TRIAL: NCT01752075
Title: A Non-interventional, Observational Post-marketing Registry of Patients Treated With Revlimid (Lenalidomide) in Taiwan
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: T-CC-5013-MM-009
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- REVLIMID: Taiwanese patients treated with REVLIMID
  Interventions: Drug: Revlimid

INTERVENTIONS:
Drug: Revlimid — The prescribing physician should prescribe and monitor REVLIMID therapy according to the guidance and recommended schedules given in the approved Taiwan package insert (PI).
  Other Names: Lenalidomide; CC-5013

SUMMARY:
The REVLIMID Registry will provide safety data from a large cohort of Taiwanese patients treated with REVLIMID. In addition, the registry will provide efficacy data and outcomes in a real-world setting (versus a clinical trial).

DETAILED DESCRIPTION:
The REVLIMID Registry is a prospective, multi-center, observational study. The registry will register 100 patients being prescribed REVLIMID in Taiwan during and patients will be followed for two years after the enrollment of the last patient.

Safety and efficacy data will be recorded in the registry monthly or bi-monthly. In accordance with the Risk Minimization Program for REVLIMID (RevAssure) a patient categorized as a woman of childbearing potential will be prescribed REVLIMID on a monthly basis, whereas women of non-childbearing potential and men will be allowed up to two months supply per prescription.

After entry of baseline data, the prescribing physician should prescribe and monitor REVLIMID therapy according to the guidance and recommended schedules given in the approved Taiwan package insert (PI)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older
* Patients that are being prescribed REVLIMID in combination with dexamethasone for the treatment of multiple myeloma and that have received at least one prior therapy
* Patient must be willing and able to provide informed consent
* Patients will be informed about the Registry and will have to sign a specific Registry Informed Consent Form
* Be able to ask questions prior to signing the Subject Information and Consent Form
* Be clearly informed that their involvement/participation in the registry is voluntary
* Understand that their medical care will not be altered in any way by their participation in the registry

Exclusion Criteria:

- A Patient who is unwilling or unable to provide informed consent will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Taiwanese patients with relapsed/refractory multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2013-07-12 (Actual); Study Completion 2013-07-19 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to two years
  Number of participants with adverse events

SECONDARY OUTCOMES:
Efficacy | Up to two years
  Revlimid dosage, reason for Revlimid discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Ye Hua, MD, Study Director — Celgene
Locations (1):
- NTUH, Taipei, Taiwan